CLINICAL TRIAL: NCT05545969
Title: A Multicentre, Open Label, Phase II Study to Determine the Response to Neoadjuvant Pembrolizumab and Lenvatinib Followed by Adjuvant Treatment With Pembrolizumab and Lenvatinib in Mucosal Melanoma
Brief Title: Neoadjuvant Pembrolizumab and Lenvatinib for Mucosal Melanoma
Acronym: Neo PeLeMM
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Melanoma Institute Australia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIA2022/442
Record Dates: First submitted 2022-09-06; First posted 2022-09-19 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Mucosal Melanoma
Keywords: Immunotherapy; VEGF inhibitor; Neoadjuvant; Adjuvant; Pembrolizumab; Lenvatinib; Pathlogical respone
MeSH Terms: interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Intervention Model Description: Multicentre, open label, clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant and Adjuvant Therapy (Experimental): Neoadjuvant pembrolizumab & lenvatinib for 6 weeks followed by definitive surgery then adjuvant pembrolizumab alone for 46 weeks
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.
  Other Names: Keytruda
Drug: Lenvatinib — Lenvatinib is an oral potent multiple RTK inhibitor that selectively inhibits VEGF receptors, VEGFR1 (FLT1), VEGFR2 (KDR), and VEGFR3 (FLT4), fibroblast growth factor receptor (FGFR1-4), platelet derived growth factor (PDGFRα), stem cell factor receptor (KIT), and rearranged during transfection (RET)
  Other Names: Lenvima

SUMMARY:
In many cancers, early stage diagnosis and early treatment offers the best chance of a prolonged recurrence free- and overall survival. Neoadjuvant immunotherapy involves administering immune checkpoint inhibitors before surgical resection in high-risk resectable disease, such as mucosal melanoma. In resectable cancers, immune checkpoint inhibitors can enhance anti-tumour immunity by exploiting a competent immune system prior to surgery. Activating antigen-specific T cells found in the primary or baseline tumour continue to exert anti-tumour effects on remaining neoplastic cells after the resection of the original tumour, potentially preventing recurrences from occurring.

In resectable mucosal melanoma, an opportunity exists to improve clinical outcomes with the addition of neoadjuvant and adjuvant systemic therapy with nivolumab and lenvatinib as an adjunct to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histologically confirmed diagnosis of fully-resectable mucosal melanoma
* Pathological ± clinical confirmation that the presenting lesion(s) does not represent metastasis from an unknown primary cutaneous or ocular melanoma
* Measurable disease per RECIST
* Availability of a newly obtained core or excisional biopsy of an affected lesion which has not been previously irradiated
* Ability to swallow and retain oral medication
* ECOG 0 - 1
* Adequate organ function per laboratory values
* Adequately controlled blood pressure with or without anti-hypertensive medications, defined as ≤ 150/90 mmHg at screening
* Anticpated life expectabcy of > 12 months.

Exclusion Criteria:

* A diagnosis of uveal or cutaneous melanoma
* A WOCBP who has a positive serum pregnancy test within 72 hours prior to starting study treatment
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor for any disease
* Prior systemic treatment for mucosal melanoma including investigational agents. Prior surgery is acceptable
* Major surgery within 3 weeks prior to first dose of lenvatinib
* Patients who have not recovered adequately from any toxicity from other permitted anti- cancer treatment regimens
* Prior radiotherapy within 2 weeks of start of study treatment
* Received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study treatment
* Patient is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* A diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior to the first dose of study treatment
* Active autoimmune disease that has required systemic treatment in the past 12 months
* Known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known central nervous system metastases and/or carcinomatous meningitis
* A history of (non-infectious) pneumonitis//interstitial lung disease that required steroids or has current pneumonitis or current interstitial lung disease
* Active infection requiring systemic therapy
* Known history of Human Immunodeficiency Virus, active Hepatitis B or C
* Has a known history of active TB
* A current diagnosis of any gastrointestinal condition that might affect the absorption of lenvatinib
* Has a pre-existing ≥ Grade 3 gastrointestinal adverse event or a non-gastrointestinal fistula
* Prolonged QT interval >480 ms
* History of, or current cardiovascular disease
* Has a history of, or a current bleeding or thrombotic disorders or patients at risk for severe haemorrhage
* Active haemoptysis
* Patients with a ≥2+ (≥100 mg/dL) proteinuria on urine dipstick testing
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study
* Has had an allogenic tissue/solid organ transplant.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2036-05 (Estimated)

PRIMARY OUTCOMES:
Change in immune cell expression of HIF1 and immune cell densities | Baseline, week 1 week 6
  Tumour and immune cell expression of HIF1a and immune cell densities will be compared between baseline and day 8 melanoma tissue biopsies.
Pathological response rate | 6 weeks
  Proportion of patients with complete absence of residual melanoma cells in the the planned resected tumour site(s) at week 6 surgery

SECONDARY OUTCOMES:
RECIST response rate | 6 weeks
  Proportion of patients with a complete or partial RECIST response; patients with no RECIST response and patients who have RECIST confirmed disease progression in the neoadjuvant period.

OTHER OUTCOMES:
PERCIST metabolic response rate | 6 weeks
  Proportion of patients with a complete metabolic resolution (complete resolution of 18F-FDG uptake within the tumour volume); partial metabolic response (reduction of a minimum of 30% in tumour SUV normalised by lean body mass [SUL]; stable metabolic response (neither CR, PR or PD) and progressive metabolic disease (an increase of 30% in tumour SUL peak or the appearance of new lesions) in the neoadjuvant period
Immune-related response criteria | 6 weeks
  Proportion of patients with a complete or partial immune related response; patients with no response and patients who have confirmed disease progression in the neoadjuvant period
Event-free survival | 10 years
  Proportion of patients with either of: progression of disease prior to surgery or which precludes surgery, local or distant disease recurrence, mucosal melanoma related death and treatment related death, whichever occurs first from the first dose of neoadjuvant treatment or from surgery (disease recurrence).
Recurrence-free survival | 10 years
  Proportion of patients who are recurrence-free at yearly time points from the date of definitive surgery and from the end of adjuvant treatment until the end of 5 years from C1D1. To include time to any recurrence, new primary disease, locoregional recurrence and distant recurrence.
Overall survival | 10 years
  Proportion of patients alive at yearly time points from the date of first neoadjuvant study treatment (C1D1) until the end of 5 years follow up.
Incidence of any treatment-emergent adverse events | 52 weeks
  * Number, grade and duration of drug related adverse events across different grades, with attribution to pembrolizumab, lenvatinib or both.
  * Number, grade and duration of drug related adverse events requiring an interruption or permanent discontinuation of pembrolizumab, lenvatinib or both.
  * The completion rate of scheduled pembrolizumab, lenvatinib or both (administered doses / scheduled doses).
Surgical outcomes | 6 weeks
  The rate of surgical complications during and following definitive surgery
Patient reported quality of life measures | 52 weeks
  The change in longitudinal quality of life individual and overall scores from baseline.
Gut microbiome influence on response outcomes | 52 weeks
  To correlate gastrointestinal mucosal integrity with bacterial composition in stool samples, clinical outcomes.
Concordance of INMC-rated pathological response with with RECIST response, PERCIST response and immune-related response crtieria. | 6 weeks
  Concordance of pathological response with RECIST response, PERCIST response and immune-related response crtieria.

CONTACTS AND LOCATIONS:
Overall Officials: Georgina Long, MBBS, PhD, Principal Investigator — Melanoma Institute Australia
Locations (1):
- Melanoma Institute Australia, Wollstonecraft, New South Wales, Australia